CLINICAL TRIAL: NCT05397093
Title: A Phase 1a/1b, Open-Label, Multicenter Study Evaluating the Safety and Feasibility of ITIL-306 in Subjects With Advanced Solid Tumors
Brief Title: ITIL-306 in Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Instil Bio (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ITIL-306-201
Record Dates: First submitted 2022-05-25; First posted 2022-05-31 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Epithelial Ovarian Cancer; Non-small Cell Lung Cancer; Renal Cell Carcinoma
Keywords: ITIL-306; Cell Therapy; Epithelial ovarian cancer (EOC); Non-small cell lung cancer (NSCLC); Renal cell carcinoma (RCC); Fallopian tube carcinoma; Tumor Infiltrating Lymphocytes; TIL; T-cell therapy; Folate receptor α (FOLR1); Anti-folate receptor α (FOLR1); Autologous Adoptive Cell Therapy; Checkpoint, PD-1 axis inhibitor; Peritoneal carcinoma; Cellular Immunotherapy; Immuno-oncology; Costimulatory antigen receptor (CoStAR)
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Carcinoma, Non-Small-Cell Lung; Carcinoma, Renal Cell; Fallopian Tube Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1a: Dose Escalation (Experimental): Various doses will be tested in participants with EOC, NSCLC and RCC.
  Interventions: Biological: ITIL-306
- Phase 1b: Expansion (Experimental): Cohort 1: Participants with epithelial ovarian cancer (EOC)
  Cohort 2: Participants with non-small cell lung cancer (NSCLC)
  Cohort 3: Participants with renal cell carcinoma (RCC)
  Interventions: Biological: ITIL-306

INTERVENTIONS:
Biological: ITIL-306 — ITIL-306 is a cell therapy product derived from a participant's own TILs and contains a unique molecule designed to increase TIL activity when it encounters FOLR1 on the tumor. A portion of the participant's tumor is surgically removed to make a personalized ITIL-306 product. Once ITIL-306 has been made, the participant is treated with 3 days of lymphodepleting chemotherapy including cyclophosphamide and fludarabine, followed by 2 days of rest then a single infusion of ITIL-306.

SUMMARY:
ITIL-306-201 is a phase 1a/1b, multicenter, clinical trial evaluating the safety and feasibility of ITIL-306 in adult participants with advanced solid tumors whose disease has progressed after standard therapy. ITIL-306 is a cell therapy derived from a participant's own tumor-infiltrating immune cells (lymphocytes; TILs) and contains a unique molecule designed to increase TIL activity when it encounters folate receptor α (FOLR1) on the tumor.

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically documented advanced (metastatic and/or unresectable) disease as appropriate per cohort.

  * Phase 1a Dose Escalation: High-grade serous epithelial carcinoma of the ovary, fallopian tube, or peritoneum, adenocarcinoma of the lung, or clear-cell renal cell carcinoma.
  * Phase 1b Expansion:

    * Cohort 1: High grade serous, endometrioid, or clear cell epithelial carcinoma of the ovary, fallopian tube, or peritoneum.
    * Cohort 2: Squamous-cell carcinoma or adenocarcinoma of the lung.
    * Cohort 3: Clear cell or papillary RCC.
* Disease must have unequivocally progressed during or after at least 1 prior line of systemic therapy that must include the following parameters (by indication):

  * Phase 1a dose escalation and Phase 1b Cohort 1: Participants with EOC whose disease has progressed during or after 1 prior line (at least 4 cycles) of platinum-based chemotherapy and had disease progression within 6 months from the last dose of the platinum agent. Participants who received 2 or more lines of platinum therapy must have disease which has progressed on or within 6 months after the date of the last dose of the platinum agent. Participants with BRCA-mutated EOC must have received previous PARP inhibitor therapy.
  * Phase 1a dose escalation and Phase 1b Cohort 2: Participants with NSCLC whose disease has progressed after 1 prior line of platinum-based doublet chemotherapy and a CPI. Participants with targetable mutations (e.g. EGFR/ALK/KRAS) are required to have progressed on targeted therapy in addition to a platinum-based doublet chemotherapy
  * Phase 1a dose escalation and Phase 1b Cohort 3: Participants with RCC whose disease has progressed after 1 prior line of antiangiogenic therapy and a PD-1-axis inhibitor.
* Medically suitable for surgical resection of tumor tissue
* Following tumor resection for TIL harvest, will have, at minimum, 1 remaining measurable lesion as identified by CT or MRI per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Adequate bone marrow and organ function

Key Exclusion Criteria:

* History of another primary malignancy within the previous 3 years
* Phase 1a:

  * EOC of the following subtypes: low-grade, endometrioid, clear cell, mucinous, sarcomatous, or mixed.
  * NSCLC of the following subtypes: squamous, neuroendocrine differentiation.
  * RCC of the following subtypes: nonclear-cell RCC
* Phase 1b:

  * Cohort 1: Participants with mucinous, sarcomatous, and low-grade EOC.
  * Cohort 2: Participants with small cell lung cancer, or NSCLC with neuroendocrine differentiation
  * Cohort 3: Participants with nonclear-cell RCC, except papillary RCC
* Previously received an allogeneic stem cell transplant or organ allograft
* Previously received TIL or engineered cell therapy (eg, CAR T-cell)
* Significant cardiac disease
* Stroke or transient ischemic attack within 12 months of enrollment
* History of significant central nervous system (CNS) disorder
* Symptomatic and/or untreated CNS metastases
* History of significant autoimmune disease within 2 years prior to enrollment
* Known history of severe, immediate hypersensitivity reaction attributed to cyclophosphamide, fludarabine, dimethyl sulfoxide (DMSO), human serum albumin (HAS), phosphate buffer or gentamycin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2022-08-24 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2039-11 (Estimated)

PRIMARY OUTCOMES:
Frequency and severity of ITIL-306 treatment-emergent adverse events (AEs), serious AEs, and AEs of special interest (AESI) | Up to 24 months

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 60 months
  ORR defined as the incidence of a complete response (CR) or a partial response (PR) per a modified Response Evaluation Criteria in Solid Tumors (RECIST v1.1) criteria, as assessed by investigator review.
Duration of response (DOR) | Up to 60 months
  For participants who experience an objective response, DOR is defined as the time from their first objective response to disease progression or death.
Progression-free survival (PFS) | Up to 60 months
  PFS is defined as the time from the ITIL-306 infusion date to the date of disease progression or death from any cause.
Overall Survival (OS) | Up to 60 months
  OS is defined as the time from the ITIL-306 infusion date to the date of death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Instil Study Director, Study Director — Instil Bio, Inc.
Locations (2):
- United States (2):
  - Washington University School of Medicine, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: No